CLINICAL TRIAL: NCT06657638
Title: Diagnostic Yield of Cytological Examination of Malignant Pleural Effusion in Different Breast Cancer Pathologies
Brief Title: Cytological Examination of Malignant Pleural Effusion in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer of chest medicine, Mansoura University Hospital
Other Study IDs: R.24.10.2828.R2
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Malignant Pleural Effusion
Keywords: malignant pleural effusion; breast cancer; Cytological examination
MeSH Terms: conditions — Pleural Effusion, Malignant; Breast Neoplasms | interventions — Thoracentesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer breast: malignant pleural effusion in breast cancer
  Interventions: Diagnostic Test: Thoracentesis

INTERVENTIONS:
Diagnostic Test: Thoracentesis — Aspiration of pleural effusion

SUMMARY:
Malignant pleural effusion (MPE) is characterized by the presence of malignant cells. It can occur in 15% of patients with cancer and is a common manifestation in patients with metastatic disease.

Breast cancer (BC) is the second most common cause of MPE and MPE occurring in 2- 11% of patients with BC. Breast cancer is a heterogeneous disease of malignant tumors with diversified morphology, clinical course, biologic behavior and prognosis, and accurate tumor classification is critical for a patient's care.

DETAILED DESCRIPTION:
The serous pleural cavity is an enclosed space covered by the parietal and visceral layers of serous membranes, which are lined by a monolayer of mesothelial cells supported on fibrous tissue rich in capillaries and lymphatic. Under physiological conditions, these two layers are in juxtaposition and only a small amount of fluid is Present inside these compartments, acting as a lubricant to avoid friction.

Many infectious, benign, and malignant diseases can cause pleural effusion. Approximately one-fourth of all pleural effusions and 30 - 70% of all exudative effusions in hospital settings are secondary to cancer.

Lung cancer is the most common metastatic tumor to the pleura in men, while breast cancer is the most common tumor in women.

Breast cancer is the most commonly diagnosed malignant tumor in women worldwide and the most common cause of malignancy- related deaths. Breast cancer patients constitute approximately 36% of all oncological patients. The incidence of breast cancer is gradually increasing worldwide.

Since breast cancer is a heterogeneous disease that varies from clinical course to molecular subtypes, it includes a wide spectrum of diseases with different presentations and morphological, biological, and clinical phenotypes. Therefore, the behavior and treatment success of breast cancer vary greatly from person to person, and, as a result, it is possible to encounter very different personalized prognosis processes in breast cancer patients.

Malignant pleural effusions are most commonly caused by carcinomas of lung, breast, gastrointestinal tract or ovary, and hematological malignancies. Diagnosis of pleural effusion is done by many maneuvers as simple aspiration for cytological examination, or using more invasive maneuvers as closed pleural biopsy and medical thoracoscopy. Large studies evaluated the sensitivity and specificity of conventional cytology for the detection of malignant cells in effusions, ranging from 40% to 80% and 89% to 98%, respectively.

Molecular classification of breast cancer was developed based on the use of complementary DNA microarrays to represent human genes. Breast cancer was divided into 4 intrinsic molecular subtypes: luminal A, luminal B, v-erb-b2 (ERBB2)/human epithelial growth factor receptor 2 (HER2) gene-overexpressing (HER2), and basal-like.

The presence of MPE in advanced cancer is associated with poor prognosis, and the range of overall survival (OS) time is from 5 to 13 months. MPE is most common in triple-negative breast cancer (TNBC), and TNBC phenotype is an unfavorable characteristic in patients with MPE, worsening the prognosis and reducing life expectancy. For symptomatic patients with MPE, it is recommended to use an indwelling pleural catheter or chemical pleurodesis combined with systemic treatment.

Several factors could be attributed to this great variability, such as different immune-cytochemical staining techniques, dilutions and type of antibody clone used, volume of sample, procedural technique and the experience of the examiner. In addition, lack of uniformity in reporting such specimens could also be a factor for such wide differences in overall values of sensitivity and specificity among studies, with no study yet, to the best of our knowledge, reporting risk of malignancy (ROM) of defined diagnostic categories in pleural fluids.

For the time being, no international recommendations have been made about the rationale of using anti-tumor therapy against standard palliative MPE treatment procedures. The clinical treatment response of MPE is poor in systemic anti-tumor therapy in most malignant conditions. Therefore, there is an urgent need to develop a viable and reliable method to improve therapeutic effects of BC patients with MPE.

Therefore, pleural effusion samples will be sampled, using a diagnostic system and reporting ROM for each defined category, as well as use of immunohistochemistry and overall sensitivity and specificity of cytology when compared to concomitant pleural biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are presented for thoracentesis with routine cytological examination of pleural effusion before biopsy or thoracoscopy, if the appearance of visceral and parietal pleural was clearly and if malignant diagnosis of breast was confirmed on histological analysis of the biopsy material.

Exclusion Criteria:

* Age <18 years.
* Patients diagnosed with malignant pleural mesothelioma (MPM)
* Contraindication for pleurocentesis; patient refusing, coagulopathy and active skin infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cancer breast
Study Population: Patients are presented for thoracentesis with cytological examination of pleural effusion, if the appearance of visceral and parietal pleural was clearly and if malignant diagnosis of breast was confirmed on histological analysis of the biopsy material.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-10-19 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Cytological examination of pleural effusion in breast cancer ( cell/unit) | 6 months
  Diagnosis of pleural effusion by cytological examination

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Mansoura University
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt